CLINICAL TRIAL: NCT03330626
Title: VolumE maNagement Under Body Composition Monitoring in Critically Ill patientS on CRRT; Randomized-controlled Trial (VENUS Trial)
Brief Title: VolumE maNagement Under Body Composition Monitoring in Critically Ill patientS on CRRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Sejoong Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VENUS
Record Dates: First submitted 2017-07-01; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Renal Dialysis; Fluid Overload
Keywords: Fluid management; conventional method; InBody S10; CRRT
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: One is control for the patients under conventional methods (I/O based fluid monitoring). The other is case for the patients under Inbody S10 methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IO group (Active Comparator): Fluid overload will be removed in the patients who received continuous renal replacement therapy, but the amount of fluid removal are guided by the intake-output balance.
  Interventions: Other: IO group
- InBody group (Experimental): Fluid overload will be removed in the patients who received continuous renal replacement therapy, but the amount of fluid removal are guided by the bioimpedance analysis (InBody S10).
  Interventions: Device: InBody group

INTERVENTIONS:
Device: InBody group — As one of representative BIVA, it provides the patients' fluid status with more objective data such as TBW, ECW, ICW, etc.
  Arms: InBody group
Other: IO group — Fluid removal are guided by intake-output balance.
  Arms: IO group

SUMMARY:
Although monitoring fluid balance for continuous renal replacement therapy-treated patients is an important issue, most physicians usually use conventional methods such as the difference between the amount of intake and output (I & O), which is not objective way. Meanwhile, bioimpedance electrical vector analysis presents the patients' fluid status with more objective data. Thus, the investigators will investigate the clinical benefit for monitoring fluid balance when the investigators use InBody S10, one of representative bioimpedance electrical vector analysis, compared with conventional methods among the patients who need continuous renal replacement therapy.

DETAILED DESCRIPTION:
Although monitoring fluid balance for continuous renal replacement therapy-treated patients is an important issue, most physicians usually use conventional methods such as the difference between the amount of intake and output (I & O), which is not objective way.

Meanwhile, bioimpedance electrical vector analysis presents the patients' fluid status with more objective data.

Thus, the investigators will investigate the clinical benefit for monitoring fluid balance by using InBody S10 (0, 1, 2-day, and 7-day from CRRT initiation), one of representative bioimpedance electrical vector analysis, compared with conventional methods among the patients who need continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for INCLUSION in the study if ALL the following criteria are met;

  1. The treating clinician believes that the patient requires continuous renal replacement therapy for acute renal failure.
  2. The treating clinicians anticipate treating the patient with continuous renal replacement therapy for at least 72 hours.
  3. Informed consent has been obtained.
  4. The patient fulfills ONE of the following clinical criteria for initiating continuous renal replacement therapy:

     urine output < 100 ml/6 hr that has been unresponsive to fluid resuscitation measures
     * K+> 6.5 mmol/L
     * pH < 7.2
     * Urea > 25 mmol/L
     * Clinically significant organ edema in the setting of acute kidney injury
  5. Patients who are over 5% of fluid overload or their total body water/height^2 ≥13 L/m^2

     Exclusion Criteria:
* Patients will be EXCLUDED from the study if, in the opinion or knowledge of the responsible clinician ANY of the following criteria are present:

  1. Patient age is < 18 years
  2. Death is imminent (<24 hours)
  3. There is a strong likelihood that the study treatment will not be continued in accordance with the study protocol.
  4. The patient has been treated with continuous renal replacement therapy or other dialysis previously during the same hospital admission.
  5. The patient has been on maintenance dialysis prior to the current hospitalization.
  6. Any other major illness that, in the investigator's judgement, will substantially increase the risk associated with the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate reaching euvolemia | 7 days from CRRT initiation
  To compare how many rates the two groups reach the euvolemia at 7 days from CRRT initiation

SECONDARY OUTCOMES:
Clinical outcomes (28-, 60-, 90-day mortality) | 28-, 60-, or 90-days
  To compare the mortality rates between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sejoong Kim, MD,PhD, Principal Investigator — Department of Internal Medicine, Bundang Seoul National University Hospital
Locations (1):
- Bundang Seoul National University Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Oh HJ, An JN, Oh S, Rhee H, Lee JP, Kim DK, Ryu DR, Kim S. VolumE maNagement Under body composition monitoring in critically ill patientS on CRRT: study protocol for a randomized controlled trial (VENUS trial). Trials. 2018 Dec 12;19(1):681. doi: 10.1186/s13063-018-3056-y. PMID 30541593